CLINICAL TRIAL: NCT05281328
Title: A Randomized, Placebo-controlled, Double-blind, Multi-center Trial to Assess Efficacy and Safety of Octreotide Subcutaneous Depot (CAM2029) in Patients With Symptomatic Polycystic Liver Disease
Brief Title: A Trial to Assess the Efficacy and Safety of Octreotide Subcutaneous Depot in Patients With PLD
Acronym: POSITANO
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Camurus AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HS-20-677; 2021-003764-27 (EudraCT Number)
Record Dates: First submitted 2022-03-07; First posted 2022-03-16 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Polycystic Liver Disease
Keywords: Polycystic liver; PLD; ADPLD; ADPKD; PCLD; height-adjusted total liver volume; htTLV; CAM2029; POSITANO
MeSH Terms: conditions — Polycystic liver disease; Polycystic Kidney, Autosomal Dominant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- CAM2029 once weekly (Experimental): 0.5 mL CAM2029 10 mg, subcutaneous (SC) injection, once weekly
  Interventions: Drug: CAM2029
- CAM2029 once every 2 weeks (Experimental): 0.5 mL CAM2029 10 mg, SC injection, every 2 weeks and 0.5 mL placebo, SC injection, once every 2 weeks (alternating with CAM2029 dosing)
  Interventions: Drug: CAM2029; Drug: Placebo
- Placebo (Placebo Comparator): 0.5 mL placebo, SC injection, once weekly
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CAM2029 — SC injection using a pre-filled pen
  Other Names: octreotide subcutaneous depot
  Arms: CAM2029 once every 2 weeks; CAM2029 once weekly
Drug: Placebo — SC injection using a pre-filled pen
  Arms: CAM2029 once every 2 weeks; Placebo

SUMMARY:
The purpose of the trial is to compare the effectiveness and safety of 2 treatment regimens of CAM2029 (given weekly or every 2 weeks) to placebo in participants with symptomatic PLD, either isolated as in autosomal dominant PLD (ADPLD) or associated with autosomal dominant polycystic kidney disease (ADPKD).

In the Treatment Period of the trial, participants will be allocated at random to 1 of the 3 treatment arms in a 1:1:1 ratio. After completing the Treatment Period (53 weeks) participants may proceed to a 120-week open-label extension part of the trial and then only receive the same CAM2029 treatment.

The active ingredient in CAM2029, octreotide, is administered as a subcutaneous depot using Camurus' FluidCrystal® technology.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient, ≥18 years at screening
* Diagnosis of PLD (associated with ADPKD or isolated as in ADPLD) as defined by htTLV ≥1800 mL/m at screening
* Presence of at least 1 of the following PLD-related symptoms within 2 weeks before screening: bloating, fullness in abdomen, lack of appetite, feeling full quickly after beginning to eat, acid reflux, nausea, rib cage pain or pressure, pain in side, abdominal pain, back pain, shortness of breath after physical exertion, limited in mobility, concern about abdomen getting larger, dissatisfied by the size of abdomen
* Not a candidate for, or not willing to undergo, surgical intervention for hepatic cysts during the trial

Exclusion Criteria:

* Surgical intervention for PLD within 3 months before screening
* Treatment with a somatostatin analogue (SSA) within 3 months before screening
* Non-responsive to previous treatment of PLD with an SSA as per the Investigator's assessment
* Systematic cholelithiasis within 3 months before screening or previous medical history of cholelithiasis induced by SSAs unless treated with cholecystectomy
* Presence of extrahepatic cysts that, in the Investigator's opinion, may prevent the patient from safely participating in the trial
* Severe kidney disease, as defined by eGFR <30 mL/min/1.73^m2
* Severe liver disease defined as liver cirrhosis of Child-Pugh class C
* Any other current or prior medical condition that may interfere with the conduct of the trial or the evaluation of its results in the opinion of the Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2022-06-28 (Actual); Primary Completion 2025-02-05 (Actual); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Height-adjusted total liver volume (htTLV) | From screening until treatment week 53
  Change from baseline to Week 53 in htTLV as determined by MRI volumetry

SECONDARY OUTCOMES:
PLD symptom (PLD-S) score | From screening to week 53
  Key secondary endpoint. Change from baseline to Week 53 in the PLD-S measure score
htTLV | From screening until treatment weeks 13, 25, 77, 125 and 173
  Change from baseline in htTLV as determined by MRI volumetry
PLD-S | From screening to weeks 13, 21, 25, 39, 77, 101, 125, 149 and 173
  Change from baseline in the PLD-S measure score
Height-adjusted total kidney volume (htTKV) | From screening until treatment weeks 13, 25, 53, 77, 125 and 173
  Change from baseline in htTKV as determined by MRI volumetry
Total liver cyst volume | From screening to treatment weeks 13, 25, 53, 77, 125 and 173
  Change from baseline in total liver cyst volume determined by MRI volumetry
Estimated glomerular filtration rate (eGFR) | From treatment week 1 to weeks 13, 25, 53, 65, 77, 101, 125, 149 and 173
  Change from baseline in eGFR, assessed by the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) cystatin C equation using serum concentrations of creatinine and cystatin C
PLD impact (PLD-I) score | From screening to weeks 13, 21, 25, 39, 53, 77, 101, 125, 149 and 173
  Change from baseline in the PLD-I measure score
Clinical Global Impression of Severity (CGI-S) score | From treatment week 1 to weeks 13, 21, 25, 53, 77, 101, 125, 149 and 173
  Change from baseline in the CGI-S score
Patient Global Impression of Severity (PGI-S) score | From screening to weeks 13, 21, 25, 39, 53, 77, 101, 125, 149 and 173
  Change from baseline in the PGI-S score
Patient Global Impression of Change (PGI-C) score | At treatment weeks 13, 21, 25, 39, 53, 77, 101, 125, 149 and 173
  Change from baseline in the PGI-C score
Short Form-36 (SF-36) score | From treatment week 1 to weeks 25, 53, 77, 101, 125, 149 and 173
  Change from baseline in the SF-36 score
Polycystic Liver Disease Questionnaire (PLD-Q) | From treatment week 1 to weeks 25, 53, 77, 101, 125, 149 and 173
  Change from baseline in the PLD-Q score
Adverse events (AEs) | From screening to the safety follow-up, assessed up to approximately 43 months
  Incidence of AEs

CONTACTS AND LOCATIONS:
Overall Officials: Joost Drenth, MD, Principal Investigator — Department of Gastroenterology and Hepatology, Radboud UMC Nijmegen, The Netherlands
Locations (11):
- United States (6):
  - Mayo Clinic, Rochester, Minnesota
  - Mount Sinai Hospital, New York, New York
  - The New York Presbyterian Hospital, New York, New York
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Bon Secours Richmond Community Hospital, Richmond, Virginia
- University Hospitals KU Leuven, Leuven, Belgium
- Germany (3):
  - Hannover Medical School, Hanover
  - Universitätsklinikum Leipzig, Leipzig
  - Universitaetsklinikum Müenster, Münster
- Radboud UMC, Department of Gastroenterology and Hepatology, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] St Pierre K, Cashmore BA, Bolignano D, Zoccali C, Ruospo M, Craig JC, Strippoli GF, Mallett AJ, Green SC, Tunnicliffe DJ. Interventions for preventing the progression of autosomal dominant polycystic kidney disease. Cochrane Database Syst Rev. 2024 Oct 2;10(10):CD010294. doi: 10.1002/14651858.CD010294.pub3. PMID 39356039